CLINICAL TRIAL: NCT04120441
Title: A Fighting Chance: Pilot Study of a Group Mentoring Intervention for Assault Injured Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00218737
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-07

CONDITIONS: Violence
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group mentoring/Intervention (Experimental): Study participants randomized to intervention will be enrolled in a Y in Central Maryland group mentoring program that meets weekly over a three month period. Parents will participate in three parenting sessions. Youth study participants will be interviewed about the youth's thoughts and behaviors and the youth's medical and school records will be reviewed. Parents will also be interviewed to ask questions about the program. The study will last for 12 months and youth/parents will be interviewed at the time of enrollment and 4-6 months later.
  Interventions: Behavioral: Group Mentoring/Intervention
- Routine care/control (No Intervention): Study participants randomized to control will receive information about community resources. Youth study participants will be interviewed about the youth's thoughts and behaviors and the youth's medical and school records will be reviewed. Parents will also be interviewed to ask questions about the program. The study will last for 12 months and youth/parents will be interviewed at the time of enrollment and 4-6 months later.

INTERVENTIONS:
Behavioral: Group Mentoring/Intervention — Study participants randomized to intervention will be enrolled in a Y in Central Maryland group mentoring program that meets weekly over a three month period. Parents will participate in three parenting sessions.
  Other Names: A Fighting Chance
  Arms: Group mentoring/Intervention

SUMMARY:
This pilot study is a randomized controlled trial in which assault-injured 12-14 year old youth recruited from the emergency department (ED) are randomly assigned to standard care or "A Fighting Chance" group mentoring.

DETAILED DESCRIPTION:
The goal of this project is to adapt, implement and evaluate Take Charge! (a 1:1 mentoring intervention for assault-injured youth) for a group mentoring model.

This pilot study is a randomized controlled trial in which assault-injured 12-14 year old youth recruited from the emergency department are randomly assigned to standard care or "A Fighting Chance" group mentoring that includes a violence prevention curriculum and parent sessions. Immediately post-intervention and again at six-month follow up, youth violence-related, mental health and educational outcomes using validated measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Injury: Eligible youth have been treated in the ED for an interpersonal intentional injuries excluding child abuse, sexual abuse, sibling fights, police fights, and other domestic violence-related fights involving relatives and/or household residents. These excluded types of violence have a different set of complex dynamics and services needs requiring separate study and intervention.
* Age: Eligible youth are age 12-14 years (i.e. up to the 14th birthday) and youths' parents/guardians are age 18 years and older.
* Mental/Physical Status: Youth and parents must have the cognitive ability to participate in the intervention. Those with severe psychopathology (i.e. severe history of mental illness with multiple psychiatric hospitalizations) or inability to comprehend questions, will be excluded.
* Language: English-speaking ability of the parent and child is necessary to enable participation in the intervention, training and assessments.
* Mentorship: Eligible youth are not currently participating in a formal mentoring program.

Exclusion criteria:

Additionally, there are youth eligibility criteria set by Y in Central Maryland policies which the investigators will follow. These include:

* Residence: Youth are not eligible if residence is outside of Baltimore City.
* Custody/child protection status: Youth are not eligible if youth have a caregiver currently involved in an ongoing custody dispute or Child Protective Services investigation. Youth are not eligible if youth live somewhere other than a residential setting with parents/guardians.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of intervention participants attending > 80% of sessions | 4-6 month follow up
  For this pilot study, the main outcome measure is that of feasibility. Specifically, the investigators will assess feasibility by determining the proportion of intervention participants that attend >80% (10 or more) sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Ryan, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No